CLINICAL TRIAL: NCT07371208
Title: Multicenter, Phase II Clinical Study of Sacituzumab Tirumotecan (Sac-TMT) in Combination With KL-A167 for Neoadjuvant Treatment of Triple-Negative Breast Cancer
Acronym: ST-A-TN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Kunwei Shen, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJBC-2503; Shanghai Jiaotong University (Other: Shanghai Jiaotong University)
Record Dates: First submitted 2026-01-18; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; triple negative; Sac-TMT; SKB264; KL-A167; neoadjuvant
MeSH Terms: conditions — Breast Neoplasms | interventions — 18-O-demethylcervinomycin A2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study cohort (Experimental): treatment arm
  Interventions: Drug: SKB264

INTERVENTIONS:
Drug: SKB264 — 1) Neoadjuvant Treatment Phase Phase a: All eligible subjects will receive Sac-TMT (5 mg/kg, Day 1, every 2 weeks) combined with KL-A167 (900 mg, Day 1, every 2 weeks) for 6 cycles (12 weeks).
  At Week 12 (beginning of Week 13), radiographic assessment via contrast-enhanced breast MRI will be performed. Based on tumor response, patients proceed to Neoadjuvant Phase b:
  i. Responders (investigator-assessed Partial Response [PR] or Complete Response [CR]): Continue the same combination regimen for an additional 12 weeks of neoadjuvant therapy.
  ii. Non-responders (investigator-assessed Stable Disease [SD] or Progressive Disease [PD]): Switch to KL-A167 (900 mg every 2 weeks) combined with nab-paclitaxel (100 mg/m², Days 1, 8, 15, every 4 weeks per cycle) and carboplatin (AUC 2 mg·min/mL, Days 1, 8, 15, every 4 weeks per cycle) for 12 weeks.
  Other Names: KL-A167

SUMMARY:
This study is a multicenter phase II trial planning to enroll 40 patients with primary triple-negative breast cancer (tumor size ≥2 cm, clinical lymph node stage cN0-3, M0). Participants will receive the combination therapy of Sac-TMT and KL-A167 during the neoadjuvant treatment phase. The study aims to evaluate the efficacy and safety of Sac-TMT combined with KL-A167 as neoadjuvant treatment for triple-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years old.
* Diagnosis: Histologically and/or cytologically confirmed primary triple-negative breast cancer (TNBC) (excluding inflammatory breast cancer), meeting the criteria of tumor size ≥2 cm, clinical lymph node stage cN0 to cN3, and M0 (no distant metastasis). TNBC Definition: Immunohistochemistry (IHC) showing ER and PR <10%; HER2-negative: IHC 0 or 1+, or IHC 2+ with negative in situ hybridization (ISH).
* Tissue Sample: Availability of tumor tissue sample for biomarker testing.
* Measurable Disease: At least one measurable lesion according to RECIST v1.1 criteria. Lesions previously irradiated cannot be selected as target lesions. Subjects with only skin lesions or bone lesions are excluded.
* Performance Status: Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1 within 7 days prior to treatment initiation.
* Adequate Organ and Bone Marrow Function: Hematology: Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L; Platelet count (PLT) ≥ 80 × 10⁹/L; Hemoglobin ≥ 10 g/dL. Liver Function: Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤ 2.5 × upper limit of normal (ULN); Total bilirubin (TBIL) ≤ 1.5 × ULN. Renal Function: Creatinine clearance (Ccr) ≥ 60 mL/min (calculated using the Cockcroft-Gault formula). Coagulation: International normalized ratio (INR), activated partial thromboplastin time (APTT), and prothrombin time (PT) ≤ 1.5 × ULN. Cardiac Function: Left ventricular ejection fraction (LVEF) ≥ 55% as measured by echocardiography (ECHO) or multigated acquisition (MUGA) scan.
* Prior Treatment: No prior anti-tumor therapy for the current breast cancer.
* Contraception: Female subjects must have a negative serum pregnancy test. Female subjects of childbearing potential and male subjects with partners of childbearing potential must agree to use highly effective medically approved contraceptive methods from the time of signing the informed consent form until 6 months after the last dose of study drug.
* Informed Consent: Patients must voluntarily enroll in the study, provide written informed consent, and be able to comply with the protocol-specified visits and procedures.

Exclusion Criteria:

* Cardiovascular Disease: Baseline left ventricular ejection fraction (LVEF) < 55% assessed by echocardiography (ECHO) or multigated acquisition (MUGA) scan at screening, or any other significant cardiovascular disease, or myocardial disease classified as New York Heart Association (NYHA) Class III or IV.
* Prior Ipsilateral Breast Cancer: History of ipsilateral invasive breast cancer.
* Prior Treatment for Current Breast Cancer: Any prior chemotherapy, targeted therapy, and/or radiotherapy for the currently diagnosed breast cancer prior to enrollment.
* Prior Immune Checkpoint Inhibitor Therapy: Previous treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibodies, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* Prior TROP2/Topo I Inhibitor Therapy: Previous treatment with any TROP2-targeted therapy and/or topoisomerase I inhibitor.
* Other Malignancies: History of other active malignancies within the past 5 years, except for cured carcinoma in situ of the cervix, basal cell carcinoma of the skin, or squamous cell carcinoma of the skin.
* Clinically Significant Pulmonary Impairment: Clinically significant pulmonary impairment due to concurrent pulmonary disease, including but not limited to: Any underlying pulmonary disease (e.g., pulmonary embolism within 3 months prior to treatment, severe asthma, severe chronic obstructive pulmonary disease, restrictive lung disease, pleural effusion, etc.) Any autoimmune, connective tissue, or inflammatory disease with potential pulmonary involvement (e.g., rheumatoid arthritis, Sjögren's syndrome, sarcoidosis, etc.)
* History of pneumonectomy.
* CYP3A4 Modulators: Requirement for strong inhibitors or inducers of cytochrome P450 3A4 (CYP3A4) within 2 weeks prior to the first dose or during the study period (Concomitant use of strong CYP3A4 inhibitors or inducers is prohibited in this study; representative agents are listed in Appendix 2). All subjects must avoid concomitant use of any known CYP3A4-inducing drugs, herbal supplements, and/or food.
* Contraindications/History: Known history of allergy/hypersensitivity to the study drugs or their components; history of immunodeficiency; history of organ transplantation.
* Interstitial Lung Disease (ILD)/Pneumonitis: History of (non-infectious) interstitial lung disease (ILD) or non-infectious pneumonitis requiring systemic steroid therapy. Current ILD or non-infectious pneumonitis. Suspicious ILD or non-infectious pneumonitis on imaging at screening that cannot be ruled out by imaging evaluation.
* Ocular Diseases: Documented severe dry eye syndrome, severe meibomian gland dysfunction and/or blepharitis, or history of corneal disease that may delay corneal epithelial healing.
* Active Autoimmune Disease: Active autoimmune disease that has required systemic treatment within the past 2 years (Note: Hormone replacement therapy is not considered systemic treatment; e.g., type I diabetes, hypothyroidism managed with thyroid hormone replacement only, adrenal or pituitary insufficiency managed with physiologic corticosteroid replacement only).
* Active Infection: Active infection requiring systemic therapy within 2 weeks prior to the first dose.
* Uncontrolled Comorbidities: Any significant concurrent illness, in the investigator's judgment, that may jeopardize patient safety or affect study completion, including but not limited to uncontrolled hypertension, severe diabetes, active infection, etc.
* Investigator Discretion: Any condition that, in the investigator's opinion, could interfere with the evaluation of the study drug, compromise patient safety, or interpretation of study results, or any other condition that makes the subject unsuitable for study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-24 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
pCR | after neoadjuvant treatment, at surgery
  ypT0/Tis ypN0

SECONDARY OUTCOMES:
ORR | after neoadjuvant treatment, at surgery
  ORR per RECIST v1.1
EFS | From enrollment to 5 years after surgery
  EFS
OS | From enrollment to 5 years after surgery
  OS
Safety | through study completion, an average of 1 year
  Safety per NCI CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Jiaotong University School of Medicine affiliated Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided